CLINICAL TRIAL: NCT04320394
Title: Evaluation of Sepsis-induced Immunosuppression Base on QuantiFERON Monitor® in Patients Presenting to the Intensive Care Unit for Septic Shock
Brief Title: Evaluation of Sepsis-induced Immunosuppression Base on QuantiFERON Monitor® in Septic Shock
Acronym: MONITOR SEPSIS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-AOI-08
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2020-03

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: Monocentric, Open-Label prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Septic shock patients (Other): Patients with septic shock will be taken from an additional tube to analyze their immune response
  Interventions: Diagnostic Test: QuantiFERON Monitor®

INTERVENTIONS:
Diagnostic Test: QuantiFERON Monitor® — The test will be realised to evaluate sepsis induced immunosuppression on patient with septic shock

SUMMARY:
QuantiFERON Monitor® is an immunological test evaluating the nonspecific cellular response by measuring interferon gamma (IFNγ) secretions after T-cell and natural killer lymphocyte stimulation.

This study aims at evaluating sepsis-induced immunosuppression base on QuantiFERON Monitor® in patients presenting to the intensive care unit for septic shock. The sponsor expects to identify sepsis-induced immunodeficiency in patients through a better understanding of cellular and adaptive immune responses.

DETAILED DESCRIPTION:
A sepsis-induced immunosuppression phase has recently been characterized and has been associated with worse outcomes as well as increased healthcare costs. Furthermore, a marked suppression of the immune response has been partially described in patients hospitalized in the intensive care setting but its monitoring is not available in daily practice. QuantiFERON Monitor® is an immunological test evaluating the nonspecific cellular response by measuring interferon gamma (IFNγ) secretions after T-cell and natural killer lymphocyte stimulation. Several studies have shown the pertinence of this test, especially in patients with kidney failure requiring renal replacement therapy. Patients with lower IFNγ levels were also found to be at higher risk of infection.

This study aims at evaluating sepsis-induced immunosuppression base on QuantiFERON Monitor® in patients presenting to the intensive care unit for septic shock. The sponsor expects to identify sepsis-induced immunodeficiency in patients through a better understanding of cellular and adaptive immune responses. This should ultimately lead to determining thresholds for sepsis-related complications and identifying patients most at risk of sepsis-induced immuno-depression.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in intensive care and intensive care at Nice University Hospital and presenting with septic shock (defined by the presence of sepsis, the need for a vasopressor to maintain a MAP> 65mmHg and hyperlactatemia> 2mmol / l)
* Free and express informed consent signed by the patient or the confidential counselor in case of impossibility (deferred consent of the patient as soon as his condition allows it)
* Age> 18 years old
* Affiliated to a social security scheme

Exclusion Criteria:

* Pregnant woman Patient under the age of 18
* Patient under guardianship or curatorship or placed in detention
* Patient with congenital or previously acquired immune deficiency
* Patient on prior immunosuppressive treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
identification of patients with sepsis-induced immunosuppression in a population of patients with septic shock, by an objective and functional immunological test measuring the production of IFN-γ, the QuantiFERON Monitor® | 24 months
  Use of an objective and functional immunological test measuring the production of IFN-γ, the QuantiFERON Monitor®

SECONDARY OUTCOMES:
obtaining a threshold value of IFN - γ in the plasma of patients to define an immunosuppression threshold and then to predict the occurrence of secondary infectious complications. | 24 months
  the value of IFN - γ (UI/mL) in the plasma will be mesured after stimulation of the immune cells,

IPD SHARING:
Plan to Share IPD: No
no data sharing plan is planned